CLINICAL TRIAL: NCT04558944
Title: Clinical Use of the Extracorporeal Shock Wave Therapy in the Treatment of Pathological Post Burn Scars
Brief Title: The Effect of Extracorporeal Shock Wave Therapy in the Treatment of Post Burn Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR(ATR)398/2016
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Cicatrix, Hypertrophic
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Two randomized groups with twenty patients per group. The control group received the standard treatment for postburn scars. The treatment group (ESWT) received the standard treatment and treatment of postburn scars with ESWT 512 impulses of o.15mJ/mm 2 in each session, twice per week for 4 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This group received pain and pruritus medication as needed, received the usual physical therapy as per the protocol of our burn unit, as well as compression garments, silicone sheets and gels and moisturizing cream twice a day. Additionally, the patients were advice on reducing sun exposure and applying +50SPF sunblock on a daily basis.
- Extracorporeal Shock Wave Therapy group (Experimental): This group received the same treatment as the control group plus Extracorporeal Shock Wave Therapy (The DermaPACE® System, SANUWAVE Health Inc., USA) with Energy Flux Density of 0.15mJ/mm 2 and 512 pulses per session. A total of two sessions per week during a 4-week period.
  Interventions: Device: Extracorporal Shock Wave Therapy

INTERVENTIONS:
Device: Extracorporal Shock Wave Therapy — Acoustic high amplitude waves with Energy Flux Density of 0.15mJ/mm 2 and 512 pulses per session. A total of two sessions per week during a 4-week period.
  Arms: Extracorporeal Shock Wave Therapy group

SUMMARY:
A prospective, randomized, controlled study. The patients were divided into two groups with twenty patients per group. The control group received the standard treatment for postburn scars. The treatment group received the standard treatment and treatment of postburn scars with Extracorporeal Shock Wave Therapy 512 impulses of 0.15mJ/mm 2 in each session, twice per week for 4 weeks.

The investigators assessed the appearance of scar with the Vancouver Scar Scale (VSS), pruritus and pain with Visual Analog Scale (VAS) before the start of the treatment and at 2 weeks and 5 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertrophic post burn scars of approximately 64 cm2 surface area.

Exclusion Criteria:

* Patients younger than 18 year.
* Pregnant women.
* Having a known skin condition (e.g. psoriasis, skin cancer etc.).
* Immunosuppression.
* Hemophilia .
* Matured scars.
* Scars located above the lungs, the bowels, the gonads or electronic implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Scar appearance | 6 months from inclusion
  Scar appearance by Vancouver Scar Scale. Minimum value 0. Maximum value 13. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Scar pruritus | 6 months from inclusion
  Pruritus measured by Visual Analogue Scale. Minimum value 0. Maximum value 10. Higher scores mean a worse outcome.
Scar pain | 6 months from inclusion
  Pain measured by Visual Analogue Scale. Minimum value 0. Maximum value 10. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Aguilera Sáez, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No